CLINICAL TRIAL: NCT00643006
Title: Physical Exercise and Its Impact on Signs of Inflammation in Women With Fibromyalgia
Brief Title: Physical Exercise and Its Impact on Signs of Inflammation in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other); Västra Götalands Forskningsfond (Unknown); Reumatikerförbundet (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GAU2
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Results first posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-09

CONDITIONS: Exercise Therapy; Pain
Keywords: Fibromyalgia; Physical activity; Function; Pain; Exercise; Inflammation
MeSH Terms: conditions — Pain; Fibromyalgia; Motor Activity; Inflammation | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A. High intensive exercise (Experimental): High intensive exercise
  Interventions: Behavioral: Physical exercise
- B. Low-intensive exercise (Active Comparator): Low-to-moderate intensive supervised walks
  Interventions: Behavioral: Active comparator: low intensive exercise

INTERVENTIONS:
Behavioral: Physical exercise — Supervised walks with poles twice a week at moderate-high intensity
  Arms: A. High intensive exercise
Behavioral: Active comparator: low intensive exercise — Supervised walks once a week at low-intensity.
  Arms: B. Low-intensive exercise

SUMMARY:
The study aims to compare low-intensive and high-intensive physical exercise and its impact on physical function, pain and signs of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Women with Fibromyalgia, interested in exercise twice a week

Exclusion Criteria:

* Other severe diseases

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa E Mannerkorpi, Ass prof, Principal Investigator — Göteborg University, Dept of Rheumatology
Locations (3):
- Sweden (3):
  - Alingsås Primary Health Care, Alingsås
  - Sahlgrenska University Hospital, Dept of Physical Therapy, Gothenburg
  - Uddevalla Primary Health Care, Uddevalla

REFERENCES:
- [Derived] Bjersing JL, Erlandsson M, Bokarewa MI, Mannerkorpi K. Exercise and obesity in fibromyalgia: beneficial roles of IGF-1 and resistin? Arthritis Res Ther. 2013 Feb 27;15(1):R34. doi: 10.1186/ar4187. PMID 23446104
- [Derived] Bjersing JL, Dehlin M, Erlandsson M, Bokarewa MI, Mannerkorpi K. Changes in pain and insulin-like growth factor 1 in fibromyalgia during exercise: the involvement of cerebrospinal inflammatory factors and neuropeptides. Arthritis Res Ther. 2012 Jul 9;14(4):R162. doi: 10.1186/ar3902. PMID 22776095
- [Derived] Mannerkorpi K, Nordeman L, Cider A, Jonsson G. Does moderate-to-high intensity Nordic walking improve functional capacity and pain in fibromyalgia? A prospective randomized controlled trial. Arthritis Res Ther. 2010;12(5):R189. doi: 10.1186/ar3159. Epub 2010 Oct 13. PMID 20942911

RESULTS

PARTICIPANT FLOW:
Groups:
- A. High Intensive Exercise: High intensive exercise by means of Nordic walking twice a week for 45 minutes during 15 weeks
- B. Low-intensive Exercise: Low-to-moderate intensive supervised walks twice a week for 45 minutes during 15 weeks
Period: Overall Study
Arm/Group | A. High Intensive Exercise | B. Low-intensive Exercise
Started | 34 | 33
Completed | 29 | 29
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A. High Intensive Exercise | B. Low-intensive Exercise | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 33 | 67
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (7.8) | 50 (7.6) | 49 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Six-minute Walk Test
Description: Patient is instructed to walk as fast as she can. The distance covered during 6 minutes is documented.
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: meter
Groups:
- Arm A. Exercise: The intervention group participated in Nordic walking
- Arm B. Active Comparator: The active comparison group participated in low-intensive walks.
Arm/Group | Arm A. Exercise | Arm B. Active Comparator
Number analyzed (Participants) | 29 | 29
meter | 37.7 (41.8) | 8.6 (42.2)

2. Primary Outcome: Change of Pain Level From Baseline.
Description: Pain was measured by The Fibromyalgia Impact Questionnaire (FIQ) subscale for Pain, which is a self-rated pain on visual analogue scale, 0-100 mm. The higher value, the worse pain.
Time Frame: 15 weeks
Population: Patients attending at post-test
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | A. High Intensive Exercise | B. Low-intensive Exercise
Number analyzed (Participants) | 29 | 29
mm | -4.0 (14.5) | -5.3 (16.3)

ADVERSE EVENTS:
Arm/Group | A. High Intensive Exercise | B. Low-intensive Exercise
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No